CLINICAL TRIAL: NCT02496949
Title: A Phase Ib ,Single Center, Open-labeling, Multiple Oral Dose Study to Assess the Safety, Tolerability，PK and Efficacy Profile for Advanced Solid Tumor Patients in China
Brief Title: A Phase Ib Study to Assess Safety and Efficacy of Oral Icaritin in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing Shenogen Biomedical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Binghe Xu, Internal medicine director,Cancer institute & hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG1114ICR
Record Dates: First submitted 2015-07-05; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Solid Tumors
MeSH Terms: interventions — icaritin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Icaritin (Experimental): 600mg,800mg two doses, Bid, continuous dosing for 56 days, to assess the safety,tolerance,pharmacokinetics and efficacy of icaritin
  Interventions: Drug: Icaritin

INTERVENTIONS:
Drug: Icaritin — 600mg,800mg two doses, Bid, continuous dosing for 56 days, to assess the safety,tolerance,pharmacokinetics and efficacy of icaritin
  Other Names: IC-162

SUMMARY:
to assess the safety, tolerability，PK and efficacy profile of two doses (600mg,800mg,BID) of Icaritin in advanced solid tumor patients in China

DETAILED DESCRIPTION:
Estrogen receptor,ERa36, predominantly localizes on the plasma membrane and in the cytoplasm and mediates a membrane-initiated "nongenomic" signaling pathway. Membrane-initiated estrogen signaling has been linked to rapid responses to estrogen and generally activates signaling pathways like the mitogen-activated protein kinase/extracellular signal-regulated kinases (MAPK/ERK), phosphatidylinositol-3-kinase, and protein kinase C pathways. Preclinical study demonstrated that ERa36 was expressed in tumor cells and might be the driving force of breast cancer cell proliferation. 40% of breast cancer tumors which used to be considered as ER negative also express ERa36. In the former study the investigators found that 40% of ERa66-positive breast cancer patients express high levels of ERa36 in their tumors, and this subset of patients are less likely to benefit from tamoxifen treatment compared with those with ERa66-positive/ERa36-negative tumors.

Icaritin is a newly discovered small molecule with selective ERa36 modulating capability and the potential as a very promising new drug to treat advanced breast cancer and hepatocellular carcinoma (HCC) by targeting this nongenomic pathway. Studies showed that it can inhibit the growth of cancer cells both in vitro and in vivo. The investigators have completed the preclinical pharmacokinetic, pharmacodynamic (PK&PD) and toxicity studies in animals and now move on to test it in a phase Ib clinical trial.

ELIGIBILITY:
Inclusion criteria:

1. age≥18 years old and ≤65
2. The patients with advanced breast tumors，hepatocellular carcinoma (HCC) or other advanced solid tumor patients who are confirmed through histologic or cytologic diagnosis to be ER positive or subjects whom investigators believe may benefit from the trial.
3. Patients with advanced cancer that relapsed after or failed previous standard treatment
4. 19≤BMI index≤30
5. No serious heart, liver,lung and kidney diseases.
6. .Received at least one anti-cancer treatment (including chemotherapy, radiotherapy, biological or endocrine treatment). And the last treatment must be at least four weeks before study enrollment or after 5 times of the drug's half-life time has passed. The surgery treatment must be more than three months.
7. Life expectancy of at least 12 weeks. 8 .Patients who can cooperate to observe AE and efficacy.

9. No any other concurrent anti-cancer treatment 10. A signed informed consent must be obtained prior to performing any study specific procedures.

11. The Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 12. Female:Women with childbearing potential must have a negative pregnancy test performed 13. HCC patients: Child-Pugh Class of A or B

Exclusion Criteria:

1. Have a known hypersensitivity to flavonoid drugs.
2. Hepatic:

   1. HCC patients : ALB <2.8g/dL, TB>3.0mg/dL, ALT and AST > 2.5 times the upper limit of Normal
   2. Advanced breast tumors or other advanced solid tumor patients: ALB >limit of normal, TB> the upper limit of normal, ALT and AST > upper limit of Normal Renal: Serum Creatinine >1.5 times the upper limit of normal. Blood test: Absolute neutrophil count (ANC) < 1.5 × 109/L, Platelet count < 90 × 109/L, Hemoglobin <9 g/dL.
3. PT/APTT >1.25 times the upper limit of normal. HCC patients: PT > 5 seconds above control
4. Suffered from thrombotic disease.
5. Serum Ca > the upper limit of normal.
6. Not recovered from toxic effects of previous anti-cancer treatments or surgery.
7. Any serious or uncontrollable concomitant systemic disorder (such as unstable respiratory disorders, cardiovascular, hepatic or kidney disorders.) or active infection which will influence the clinical trial.
8. CNS metastases or invade requiring treatment for unstable status or various psychiatric disorders
9. Malabsorption or other disease which will affect the drug absorption,distribution,metabolism and excretion.
10. Other concurrent malignancies with the exception of cervical cancer in situ or squamous cell carcinoma of the skin .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The number of patients reported adverse events | 1-2 year

SECONDARY OUTCOMES:
Progression free survival | 1-2 Years
Time to tumor progression | 1-2 Years
Overall survival | 1-2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Bing he Xu, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer institute & hospital, chinese academy of medical sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Fan Y, Li S, Ding X, Yue J, Jiang J, Zhao H, Hao R, Qiu W, Liu K, Li Y, Wang S, Zheng L, Ye B, Meng K, Xu B. First-in-class immune-modulating small molecule Icaritin in advanced hepatocellular carcinoma: preliminary results of safety, durable survival and immune biomarkers. BMC Cancer. 2019 Mar 28;19(1):279. doi: 10.1186/s12885-019-5471-1. PMID 30922248